CLINICAL TRIAL: NCT01549522
Title: Phase 1 0 Qualitative Research for Stage 4 Liver Cancer Patients and Their Caregivers.
Brief Title: Qualitative Research for Stage 4 Liver Cancer Patients and Their Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Find A Cure Panel (Other)
Responsible Party: Principal Investigator, Douglas Lowell, Recruiter, Find A Cure Panel
Other Study IDs: facplc1001
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Stage 4 Liver Cancer
Keywords: patients or caregivers; for caregivers, loved one must still be living
MeSH Terms: conditions — Liver Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: bulletin board or telephone depth interview (TDI) — experiential based research. anonymous participation.
Behavioral: interview regarding experiences and opinions as to condition and treatment — not a drug trial. experential/opinion based research.

SUMMARY:
This is opinion based, experiential research and is NOT a drug trial.

ELIGIBILITY:
Inclusion Criteria:

* stage 4 liver cancer patients and caregivers

Exclusion Criteria:

* loved ones passed away

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver cancer stage 4 patients and caregivers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National, Los Angeles, California, United States

REFERENCES:
- See also: Related Info — http://www.findacurepanel.com